CLINICAL TRIAL: NCT02942069
Title: Reproducibility of Glucose Fluctuations by Standardized Exercise for Patients With Type 1 Diabetes - a Method Study Based on Continuous Glucose Monitoring
Status: Completed | Type: Observational
Sponsor: Nordsjaellands Hospital (Other)
Responsible Party: Principal Investigator, Gabriel Tafdrup Notkin, Physiotherapist, Nordsjaellands Hospital
Other Study IDs: T1DM&CGM
Record Dates: First submitted 2016-10-20; First posted 2016-10-21 (Estimated); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Diabetes Mellitus, Type 1; Exercise; Continuous Glucose Monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Blood glucose measured using CGM during standardized physical activity — Standardized exercise on bicycle at 70% of the participants work capacity for ½ hour.

SUMMARY:
The purpose of this project is to investigate whether the glucose response in type 1 diabetes patients measured using Continuous Glucose Monitoring measurement is reproducible in repeated standardized test sessions that include physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes with a diabetes duration of at least 2 years
* age 18-60 years (inclusive)
* given informed consent
* exercises (at least 30 minutes intentional exercise where participants feel exhausted) one or more times a week
* participants agree to use CGM correctly

Exclusion Criteria:

* pregnancy
* exercising at a high level (five or more times a week with high intensity)
* treatment with prednisolone or less than a month ago contestant has been treated with prednisolone
* treatment with beta blockers
* Abuse of alcohol / drugs

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 20 patients with type 1 diabetes (treated with or without insulin pump) will participate in three identical test sessions on an exercise bike. During the three test sessions, patients will be monitored by heartrate, blood glucose (obtained by lancet) and CGM. The participants will also be using a diary for registration of diet as well as exercise during the study.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2016-12; Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Blood glucose response measured with CGM | 3 identical testing sessions throughout 3 weeks
  The participants will be tested on the research facility on a hospital in Denmark

CONTACTS AND LOCATIONS:
Overall Officials: Stig Mølsted, Post. doc., Study Chair — Senior Researcher
Locations (1):
- Nordsjællands Hospital, Hillerød, Denmark

IPD SHARING:
Plan to Share IPD: Yes